CLINICAL TRIAL: NCT06039774
Title: Clinical Efficacy of α-Mangostin Hydrogel Film With Chitosan Alginate Base for Recurrent Aphthous Stomatitis (RAS) Treatment
Brief Title: α-Mangostin Hydrogel Film With Chitosan Alginate Base for Recurrent Aphthous Stomatitis (RAS)
Acronym: AM-RAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pharm-202309.01
Record Dates: First submitted 2023-09-04; First posted 2023-09-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Aphthous Stomatitis
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- α-Mangostin Hydrogel Film With Chitosan Alginate Base (Experimental): Subjects will receive α-Mangostin Hydrogel Film With Chitosan Alginate Base in the form of a patch. Subjects will apply the patch once a day after breakfast or at night before sleep, subjects will be told to avoid drinking or eating for 1 hour after using the hydrogel film because these activities can remove the hydrogel film. Ulcer size and VAS score will recorded on the first day (baseline), the 3rd day, the 5th day, and the 7th day
  Interventions: Drug: α-Mangostin Hydrogel Film With Chitosan Alginate Base
- Placebo (Placebo Comparator): Subjects will receive Hydrogel Film With Chitosan Alginate Base without an active compound in the form of a patch. Subjects will apply the patch once a day after breakfast or at night before sleep and will be told to avoid drinking or eating for 1 hour after using the hydrogel film because these activities can remove the hydrogel film. Ulcer size and VAS score will recorded on the first day (baseline), the 3rd day, the 5th day, and the 7th day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: α-Mangostin Hydrogel Film With Chitosan Alginate Base — Patients will apply α-Mangostin Hydrogel Film With Chitosan Alginate Base once a day for 7 days
  Arms: α-Mangostin Hydrogel Film With Chitosan Alginate Base
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Recurrent Aphthous Stomatitis (RAS) is experienced by almost everyone and appears suddenly. Even though the risk of death due to the condition is small, its presence can make a person feel uncomfortable eating, drinking, and talking so there will be a decrease in the quality of a person's life in their daily lives. Recently, α-Mangostin (α-M) from mangosteen rind (Garcinia mangostana L) has been shown its effect to reduce oral mucosal sores on RAS in preclinical studies in rats. Therefore, research is needed to prove the benefits (efficacy) and safety of therapy in the form of a hydrogel film patch/plaster film with a chitosan alginate base as a carrier for α-Mangostin for the treatment of RAS patients.

DETAILED DESCRIPTION:
Topical medications are the primary option for addressing RAS (Recurrent Aphthous Stomatitis) due to their affordability, effectiveness, and safety. These treatments encompass various forms such as mouthwashes, aerosols, lozenges, and ointments, available in liquid, solid, and semi-solid preparations. However, employing topical drugs faces challenges related to achieving desired therapeutic outcomes. A significant hurdle is the hindered delivery of drugs to the oral mucosa, often referred to as "saliva wash out," which leads to the removal and rinsing away of the drug from the mucosal surface.

Efforts in developing drug delivery systems for RAS treatment are directed towards achieving several goals. These include prolonging the time drugs remain effective at the site of the ulcer, ensuring the release of adequate drug concentrations to the ulcer, and alleviating pain. Addressing this issue involves the creation of film formulations that can serve as a protective layer for the ulcer. Such formulations act as barriers against external stimuli while offering a certain degree of pain relief.

An indigenous plant of Indonesia that has found application in traditional healing is the mangostin peel (Garcinia mangostana L.). α-mangostin, extracted from the rind of the mangosteen, has been employed in traditional medicine. Among its attributes, α-mangostin exhibits anti-inflammatory properties, functioning effectively by impeding the inflammatory response. This characteristic positions α-mangostin as a viable alternative compound for addressing RAS management. To facilitate the delivery of α-mangostin, a combination of two mucoadhesive polymers, specifically sodium alginate and chitosan, is utilized as a drug delivery system.

In earlier studies, the development and analysis of a hydrogel film containing α-mangostin, utilizing a chitosan-alginate foundation, were conducted to explore their potential for treating RAS in vivo. These experiments involved testing on white Wistar rats, resulting in a remarkable 93% healing rate by the seventh day. Consequently, additional research focusing on the chitosan-alginate based α-mangostin hydrogel film will progress to clinical and safety trials. The objective is to establish its effectiveness among RAS patients and assess its suitability as a readily applicable treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-59years
* Healthy subjects without mouth diseases
* Not using drugs for RAS therapy
* Not involved with other clinical trials
* Willing to participate

Exclusion Criteria:

* Have a mouth disease
* Have other serious illnesses, including arrhythmia, uncontrolled hypertension, diabetes, hepatitis, and kidney failure
* pregnant or lactating women, and women who wish to become pregnant during the study period
* poor oral hygiene that requires treatment
* chronic diseases requiring treatment with antibiotics, hormones, nonsteroidal anti-inflammatory drugs, immunosuppressants, immune enhancers, cytotoxic drugs, or cell cycle agents that affect the oral mucosa
* mental illness or limited mental capacities

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-04 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Ulcer Size | 7 days
  The diameter of the ulcer will be measured twice (day 1 and day 7) using a ruler.
Pain Visual Analogue Scale (VAS Score) | 7 days
  Determine the effect of α-Mangostin for reducing pain intensity. The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 (no pain) and 10 (the worst pain ever felt / imagined by the subject). After being explained, subjects will be asked to place a mark on the line to rate their current level of pain. The investigators will measure the distance of the mark from 0 end point using a ruler and record the number up to 1 decimal point.
  VAS scores will be measured and recorded twice, i.e. day 1 and day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Indah Suasani Wahyuni, drg., Principal Investigator — Faculty of Dentistry Universitas Padjadjaran Bandung
Locations (1):
- Padjadjaran University Dental and Oral Hospital, Bandung, West Java, Indonesia

REFERENCES:
- [Derived] Vitamia C, Iftinan GN, Latarissa IR, Wilar G, Cahyanto A, Mohammed AFA, El-Rayyes A, Wathoni N. alpha-Mangostin hydrogel film with chitosan alginate base for recurrent aphthous stomatitis (RAS) treatment: study protocol for double-blind randomized controlled trial. Front Pharmacol. 2024 Feb 16;15:1353503. doi: 10.3389/fphar.2024.1353503. eCollection 2024. PMID 38434698